CLINICAL TRIAL: NCT00615355
Title: Efficacy of Narrow-band UVB Treatment After Transplantation of Harvested Epidermal Cells in Vitiligo
Brief Title: Epidermal Cell Transplantation in Vitiligo Skin With and Without Narrow-band Ultraviolet B (UVB) Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 18-262 ex 06/07
Record Dates: First submitted 2008-02-02; First posted 2008-02-14 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Vitiligo
Keywords: vitiligo; narrow-band UVB; ReCell; transplantation; laser
MeSH Terms: conditions — Vitiligo | interventions — Radiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body location (Other): Different body locations receive specific treatments
  Interventions: Radiation: UVB 311 nm radiation
- Control (Active Comparator): Treatment with narrow-band UVB
  Interventions: Radiation: UVB 311 nm radiation; Device: UVB 311nm

INTERVENTIONS:
Radiation: UVB 311 nm radiation — UVB 311 nm radiation randomized to one half of the transplanted vitiligo lesion given 2 times a week for 3 months; the other half of the transplanted lesion remains UV-non-irradiated
  Other Names: narrow-band UVB
Device: UVB 311nm — Repeated UVB 311nm narrowband irradiation (24 exposures)
  Arms: Control

SUMMARY:
The effect of treatment with narrow-band UVB 311 nm after transplantation of harvested autologous epidermal cells on vitiligo lesions will be investigated.

DETAILED DESCRIPTION:
Introduction: Surgical interventions in vitiligo are widely used and additional UV exposure is often recommended after successful transplantation. However, little is known about the additional efficacy of (narrow-band) UVB due to missing comparative studies.

Aim of the study: To perform a prospective, controlled, randomized, intra-individual comparative study in vitiligo lesions treated with epidermal cell transplantation using the ReCell method with and without additional narrow-band UVB treatment.

Study design: Two weeks after transplantation of epidermal cells, one randomly chosen half of the transplanted patch will be additionally treated with narrow-band UVB therapy whereas the other half will be left untreated. For control purpose, 2 additional patches (or the two halfs of one patch) will be selected to be treated with either laser dermabrasion and narrow-band UVB or narrow-band UVB treatment alone.

Grafting with the ReCell method: A superficial skin shaving excision of 2 x 2 cm will be obtained from pigmented skin (UVA irradiation 4 weeks before the excision) using a Silver knife. A cell suspension will be obtained using the ReCell transplantation kit, according to the instructions of the manufactures. The vitiligo skin will be dermabraded by Erbium: Yag laser after local anaesthesia. Thereafter the cell suspension will be sprayed on the dermabraded skin area and fixed with special wound dressings.

Narrow-band UVB treatment: The initial UVB dose will be 50% of the minimal erythema dose, tested next to the vitiligo lesions to be treated. Treatment will be performed 2 times a week with a targeted UVB device (Dualight, TheraLight). Dose increments will be 30 mJ/cm2 at each treatment up to a dose that induces slight erythema longer than 24 hours. If this dose is reached, the dose will be reduced to the last well tolerated dose and no further increments will follow. Narrow-band UVB treatment will be performed for at least 3 months or 24 treatments.

Evaluation of the treatment success: The grade of pigmentation in all lesions will be evaluated clinically, with photographs and with laser scanning microscope every 3 weeks during the first 3 months of the study and later every 3 months within the first year. The clinical rating will be performed as follows: 0 = no repigmentation; 1 = 1-25% repigmentation; 2 = 26 to 50% repigmentation; 3 = 51 to 75% repigmentation; and 4 = 76 to 100% repigmentation. The evaluation of the photographs and the laser scanning microscopy pictures will be performed blinded by physicians not engaged in the treatment phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* 11 female or male vitiligo patients between the age of 18 and 70
* Stable vitiligo for at least 1 year

Exclusion Criteria:

* Progressive disease within the last 12 months
* Sporadic repigmentation of single patches within the last 12 months
* Patients with contraindications for UV-treatment
* Patients with anticoagulant treatment, bleeding disorders
* Patients with prolonged wound healing in the history
* History of hypertrophic scarring or keloids or Köbner phenomenon
* Reduced general health status
* Patients with allergic reactions to local anaesthesia
* Topical steroids or calcineurin inhibitors in the last 4 weeks before study entry
* UV exposure in the last 4 weeks before study entry
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
percentage of repigmentation | 3 and 6 months after transplantation

SECONDARY OUTCOMES:
stability of the achieved repigmentation | one year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Angelika Hofer, Principal Investigator — Medical Univsersity of Graz, Department of Dermatology, Austria
Locations (1):
- Medical University, Department of Dermatology, Graz, Austria